CLINICAL TRIAL: NCT04938297
Title: Rituximab,Zanubrutinib in Combination With Lenalidomide, Followed by Zanubrutinib or Lenalidomide Maintenance in Patients With Primary or Secondary CNS Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, zhoukeshu, Associate Director of Hematology, Henan Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZR2 for PCNSL/SCNSL
Record Dates: First submitted 2021-06-02; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Central Nervous System Lymphoma
Keywords: Primary CNS Lymphoma; Zanubrutinib; Lenalidomide; Rituximab; Secondary CNS Lymphoma
MeSH Terms: interventions — Rituximab; Lenalidomide; zanubrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primary CNS Lymphoma，age>65 (Experimental): 8 cycles of induction ZR2 , followed by Zanubrutinib or Lenalidomide maintenance for CR/PR fit patients through randomization by 1:1 ration
  Interventions: Drug: Rituximab, Lenalidomide, Zanubrutinib; Drug: Lenalidomide, Zanubrutinib
- Recurrent/refractory primary CNS lymphoma (Experimental): 8 cycles of induction ZR2, followed by Lenalidomide maintenance for CR/PR fit patients.
  Interventions: Drug: Rituximab, Lenalidomide, Zanubrutinib; Drug: Lenalidomide
- Recurrent/refractory diffuse large B-cell lymphoma with CNS invasion (Experimental): 8 cycles of induction ZR2, followed by Lenalidomide maintenance for CR/PR fit patients.
  Interventions: Drug: Rituximab, Lenalidomide, Zanubrutinib; Drug: Lenalidomide

INTERVENTIONS:
Drug: Rituximab, Lenalidomide, Zanubrutinib — Induction therapy: Rituximab 375 mg / m2, day 1, Zanubrutinib 160 mg bid, orally, Lenalidomide 25mg QD, orally on day 1-21, 28 days as a course of treatment, 8 courses of treatment.
Drug: Lenalidomide, Zanubrutinib — Maintenance therapy: Lenalidomide: 25mg qd (adjusted according to hectogram condition) or Zanubrutinib 160 mg bid. Continuously use for 2 years or until disease progression
  Arms: Primary CNS Lymphoma，age>65
Drug: Lenalidomide — Maintenance therapy: Lenalidomide: 25mg qd (adjusted according to hectogram condition) . Continuously use for 2 years or until disease progression
  Arms: Recurrent/refractory diffuse large B-cell lymphoma with CNS invasion; Recurrent/refractory primary CNS lymphoma

SUMMARY:
In view of the synergistic effects of rituximab, zanubrutinib, and lenalidomide and severe complications caused by current standard chemotherapy regimens in Patients for primary or secondary CNS lymphoma, we intend to conduct a prospective clinical study to evaluate the efficacy and toxicity of Rituximab, Zanubrutinib in combination with Lenalidomide. Besides, the efficacy of Zanubrutinib or Lenalidomide in maintenance was also compared.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily participate in clinical research, fully understand the study and sign the informed consent form (ICF), willing to follow and be able to complete all research steps
* histologically confirmed diffuse large B-cell lymphoma (DLBCL), all subjects must provide enough archived or fresh tumor tissue samples for immunhistochemistry (IHC) and gene expression profile (GEP) evaluation
* For untreated primary CNS lymphoma, patients should be with an age of 65 years or older, intolerable to first-line treatment
* Recurrent or refractory disease was defined as: 1) recurrence of disease after complete remission (CR), or 2) partial remission (PR), stable disease (SD), or progressive disease (PD) at the time of completion of treatment before inclusion
* Recurrent / refractory diffuse large B-cell lymphoma with CNS involvement confirmed by histopathology or imaging
* Age ≥ 18 years, ECoG score ≤ 2, expected survival time is more than 3 months
* Patients with solid lesions must obtain clear evidence of disease progression through imaging examination (head MRI or head CT) 21 days before enrollment. For patients with leptomeningeal involvement only, CSF cytology examination must confirm lymphoma cells and / or imaging findings consistent with CSF disease 21 days before enrollment (at the discretion of the investigator)
* With sufficient organ and bone marrow function , and no severe hematopoietic, heart, lung, liver, kidney, thyroid dysfunction and immune deficiency
* at least 100 days after transplantation for recurrent patients after ATST

Exclusion Criteria:

* Histologically transformed large cell lymphoma
* History of previous transplantation of allogeneic stem cells
* Received BTKi or Lenalidomide
* Received corticosteroid within 7 days for antitumor treatment
* Received chemotherapy, radiotherapy, monoclonal antibody, experimental treatment, or traditional Chinese Medicine within 4 weeks
* Received major surgery within 4 weeks
* Active malignant diseases within 2 years before entering the study
* Clinically significant cardiovascular diseases
* History of severe bleeding diseases
* history of stroke or intracranial hemorrhage within 6 months before the first administration
* Unable to swallow capsules or have diseases that significantly affect gastrointestinal function
* Uncontrolled systemic infection requiring parenteral anti infective therapy
* HIV infection or indicate active hepatitis B or C virus infection
* Drug allergies or metabolic disorders
* Pregnant or lactating women
* Any life-threatening diseases, medical conditions or organ system dysfunction that the researchers believe may affect the safety of the subjects or lead to research risks
* Required to continuously treated with potent and moderate CYP3A inhibitors or inducers
* History of deep venous thrombosis (DVT) or pulmonary embolism (PE) in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | at the end of 8 cycles of induction therapy (each cycle is 28 days)
  To evaluate the overall response rate of ZR2 in the treatment of CNS Lymphoma

SECONDARY OUTCOMES:
Overall response rate | at the end of 4 cycles of induction therapy (each cycle is 28 days) and 1 year of maintenance therapy
Progression-free survival (PFS) rate | at the end of 8 cycles of induction therapy (each cycle is 28 days), 1 year and 2 year of maintenance therapy
Overall survival（OS）rate | at the end of 8 cycles of induction therapy (each cycle is 28 days), 1 year and 2 year of maintenance therapy
Treatment related adverse events | at the end of 8 cycles of induction therapy (each cycle is 28 days), 1 year and 2 year of maintenance therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No